CLINICAL TRIAL: NCT06013020
Title: Safety and Efficacy of Century Clot-Guided Prophylactic Rivaroxaban Therapy for Post ST-Segment Elevation Myocardial Infarction Complicating Left Ventricular Thrombus Compared With Conventional Antiplatelet Therapy
Brief Title: Century Clot-Guided Prophylactic Rivaroxaban for Post STEMI Complicating Left Ventricular Thrombus
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Zunyi Medical College (Other)
Responsible Party: Principal Investigator, Cai De Jin, MD, Principal Investigator, Zunyi Medical College
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: PREVENT
Record Dates: First submitted 2023-02-28; First posted 2023-08-28 (Actual); Last update posted 2024-03-19 (Actual); Status verified 2024-03

CONDITIONS: STEMI - ST Elevation Myocardial Infarction
Keywords: Century Clot analyzer; Prophylactic; Rivaroxaban; LVT; STEMI
MeSH Terms: conditions — ST Elevation Myocardial Infarction | interventions — Rivaroxaban; Ticagrelor; Clopidogrel; Aspirin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Guided NOAC and DAPT (Experimental): The first month: rivaroxaban 2.5 mg twice daily (if CR≥24) plus standard DAPT (ticagrelor 90 mg twice daily or clopidogrel 75 mg daily plus aspirin 100 mg daily).
  The following 11 months: lower-dose ticagrelor 60 mg twice daily (45 mg twice daily if <50 kg, ≥75 yrs) or clopidogrel (75 mg daily) plus aspirin (100 mg daily).
  Interventions: Drug: NOAC+DAPT
- Unguided DAPT (Experimental): The first month: standard DAPT. The following 11 months: lower-dose ticagrelor or clopidogrel plus aspirin.
  Interventions: Drug: DAPT

INTERVENTIONS:
Drug: NOAC+DAPT — Century Clot-guided rivaroxaban plus DAPT.
  Other Names: Rivaroxaban + ticagrelor or clopidogrel + aspirin
  Arms: Guided NOAC and DAPT
Drug: DAPT — Standard DAPT for 1 month, following lower-dose ticagrelor or clopidogrel plus aspirin for 11 months.
  Other Names: Ticagrelor or clopidogrel + aspirin
  Arms: Unguided DAPT

SUMMARY:
To manage the ST-segment elevation myocardial infarction (STEMI) caused by plaque rupture, triggers platelet activation/aggregation and thrombin generation, requires dual (platelet and coagulation) pathway inhibition. However, triple antithrombotic therapy with standard dual antiplatelet therapy (DAPT) and oral anticoagulant (OAC) in the STEMI setting is a challenge, since that increase in potential risk of bleeding.

Although the incidence of left ventricular thrombus (LVT) formation after STEMI decreased in modern reperfusion therapy, including primary percutaneous coronary intervention (PCI), remains at 4% to 26%, especially that complicated by anterior STEMI. The recommendation of an OAC prophylactic therapy for preventing LVT formation in current STEMI guidelines is limited. How to optimize antithrombotic therapy to balance the bleeding-thrombotic profile, and prevent LVT formation is challenging, since insufficient evidence is available from randomized trials.

Century Clot analyzer is point-of-care testing that could assess the coagulate state: normal, hypo-coagulable, or hyper-coagulable states according to clot rate (CR) value. Whether Century Clot-guided rivaroxaban prophylactic therapy (2.5 mg twice daily, if the hypercoagulable state, defined as CR ≥24) in combination with standard DAPT could reduce LVT formation without increasing major bleeding is uncertain.

DETAILED DESCRIPTION:
The Prophylactic Rivaroxaban Therapy for Post STEMI Complicating Left VENtricular Thrombus (PREVENT) study is designed to investigate the safety and efficacy of Century Clot-guided additional low-dose rivaroxaban plus DAPT as an optimal antithrombotic strategy for preventing LVT formation after anterior STEMI undergoing primary PCI.

All eligible STEMI patients will be received standard DAPT (ticagrelor or clopidogrel plus aspirin). At post-PCI 12-24 hours, to be randomly assigned into Century Clot (CR)-guided rivaroxaban (2.5 mg twice daily for 1 month) in combination with DAPT and standard DAPT. Omitting rivaroxaban at post-PCI 1 month, and both groups are following a tailored-ticagrelor with dose reduction strategy (60 mg bid, or 45 mg bid if <50 kg, ≥75 yrs) or clopidogrel (75 mg qd) plus aspirin (100 mg qd) for further 11 months. The clinical outcome is the incidence of LVT formation, and net adverse clinical events (NACEs, composite of cardiac death, non-fatal myocardial infarction, TVR/TLR, stroke, and major bleeding) at post-STEMI 1 month, as well as at 12-month clinical follow-ups.

In PREVENT study, the investigators hypothesize that Century Clot (CR)-guided additional rivaroxaban prophylactic therapy could reduce LVT formation without increasing bleeding after anterior STEMI, when compared with standard DAPT.

ELIGIBILITY:
Inclusion Criteria:

* Ischemic chest discomfort for at least 30 minutes, with at least 1-mm (0.1-mv) ST-segment elevation in anterior leads on a standard 12-lead electrocardiogram.
* Patients provide written informed consent prior to enrollment.

Exclusion Criteria:

* Intracranial, gastrointestinal, or urogenital bleeding within 6 months
* Requiring OAC therapy (eg, atrial fibrillation, deep vein thrombosis, pulmonary thromboembolism);
* Bleeding diathesis, thrombocytopenia (platelet <100,000/mL) or hemoglobin <10 g/dL, and CRUSADE score-based high bleeding risk
* Hepatic dysfunction (serum liver enzyme>3 times the normal limit)
* Renal failure (eGFR <15 ml/min/1.73m2 or requiring dialysis)
* Severe chronic obstructive pulmonary disease
* Severe bradycardia (sick sinus syndrome or high degree atrioventricular block without pacemaker protection)
* Drugs interfering with CYP3A4 metabolism (to avoid interaction with ticagrelor): ketoconazole, itraconazole, voriconazole, clarithromycin, nefazodone, ritonavir, saquinavir, nelfinavir, indinavir, atazanavir, and telithromycin
* Life expectancy < 1 year

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 374 (Estimated)
Dates: Start 2024-04-01 (Estimated); Primary Completion 2026-12-31 (Estimated); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
The incidence of left ventricular thrombus (LVT) formation. | At 1 month
  Efficacy endpoint
The incidence of clinically significant bleeding according to International Society on Thrombosis and Hemostasis (ISTH) criteria. | At 1 month
  Safety endpoint

SECONDARY OUTCOMES:
NACE (net adverse clinical event) | At 12 months
  The incidence of NACE, including cardiac death, non-fatal myocardial infarction, target vessel/lesion revascularization, LVT formation, systemic embolism or stroke, and major bleeding.

CONTACTS AND LOCATIONS:
Overall Officials: Cai De Jin, MD, Principal Investigator — Zunyi Medical College
Locations (1):
- Affiliated Hospital of Zunyi Medical University, Zunyi, Guizhou, China

REFERENCES:
- [Background] Camaj A, Fuster V, Giustino G, Bienstock SW, Sternheim D, Mehran R, Dangas GD, Kini A, Sharma SK, Halperin J, Dweck MR, Goldman ME. Left Ventricular Thrombus Following Acute Myocardial Infarction: JACC State-of-the-Art Review. J Am Coll Cardiol. 2022 Mar 15;79(10):1010-1022. doi: 10.1016/j.jacc.2022.01.011. PMID 35272796
- [Background] Weitz JI, Angiolillo DJ, Geisler T, Heitmeier S. Dual Pathway Inhibition for Vascular Protection in Patients with Atherosclerotic Disease: Rationale and Review of the Evidence. Thromb Haemost. 2020 Aug;120(8):1147-1158. doi: 10.1055/s-0040-1713376. Epub 2020 Jun 28. PMID 32594508
- [Background] Yang WX, Lai CL, Chen FH, Wang JR, Ji YR, Wang DX. The value of Sonoclot detection technology to guide the clinical medication of the perioperative anticoagulation and antiplatelet therapy in patients with acute myocardial infarction undergoing emergent PCI. Exp Ther Med. 2017 Jun;13(6):2917-2921. doi: 10.3892/etm.2017.4336. Epub 2017 Apr 13. PMID 28587360